CLINICAL TRIAL: NCT04205747
Title: Department of Psychiatry University of Medicine and Pharmacy at Ho Chi Minh City
Brief Title: Validity and Reliability of Vietnamese Version of 17items-Hamilton Depression Rating Scale
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Nguyen Dao Uyen Trang, Resident doctor of Psychiatry, University of Medicine and Pharmacy at Ho Chi Minh City
Other Study IDs: 3697/QD-ĐHYD
Record Dates: First submitted 2019-12-18; First posted 2019-12-19 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Depression, Unipolar
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
this reseach examines the reliability and validity of 17 items- Hamilton Depression rating scale in Vietnamese population, which has been commonly used in clinical depression practice and study.

DETAILED DESCRIPTION:
- Cross-sectional study

ELIGIBILITY:
Inclusion Criteria:

* patients accept paticipating in reasearch

Exclusion Criteria:

* patients don't answer full HRDS

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients are diagnosied depressive disorder at Psychiatric and neurologic department at Unoversity of medicine and pharmacy Hochiminh city hospital
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
validity and reliability of Vietnamese version of HDRS -17 | 2020-2021
  the study measures validity and reliability of Vietnamese version of HDRS -17